CLINICAL TRIAL: NCT05968950
Title: Ultrasound Localization in Thoracic Surgery - is Radiation Reduction Achievable?
Acronym: ULTRRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bolem Nagarjun, Associate Consultant, Division of Neurosurgery, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A096602
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Thoracic Spine Disorder

STUDY DESIGN:
Intervention Model Description: Prospective, cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thoracic spine ultrasound localization (Experimental): Single arm where patients undergo both types of skin localization Experimental ( Ultrasound ) correlating with standard of care which is Thoracic spine fluoroscopy
  Interventions: Device: Thoracic ultrasound

INTERVENTIONS:
Device: Thoracic ultrasound — The use of ultrasound to count ribs in order to surface mark the corresponding spinal level

SUMMARY:
The goal of this clinical trial is to see if the investigators can find a safer and quicker way to localize the correct spinal level before the start of thoracic spinal surgery.

Currently, this localization is done with the help of spinal needles and fluoroscopy. There are some inherent issues with accuracy due to individual factors such as the type of operating table or the body habitus.

The investigators want to know if the use of ultrasound to count ribs and mark the corresponding spinal level would be a quicker and possibly even more accurate than the use of fluoroscopy.

Participants who will be approached for this study are those that have already consented to undergo thoracic spinal surgery. Once they have been consented for the study, they will undergo anesthesia as per normal and positioned prone for the intended surgery.

At this juncture, the radiographers will be setting up to perform fluoroscopy to confirm the spinal level and for the surgeons to mark the skin. For the purposes of the study, the investigators will use the ultrasound to count the ribs and mark the corresponding spinal level.

Participants will undergo fluoroscopy to mark the skin level as well. The investigators are studying to see if the ultrasound method is just as accurate as the traditional fluoroscopy method. The results will be binary and will be recorded. The study ends at this point and no further participation is required from the patient.

DETAILED DESCRIPTION:
Background & Rationale

Preoperative localization using spinal needles and fluoroscopy is the conventional method of performing the level check prior to the start of the surgery, with variations including the insertion of radio-opaque markers utilized in some units. Spinal needles are placed either over the skin or inserted directly into the body prior to taking an xray to confirm that the correct spinal levels are identified. The appropriate levels are marked on the skin and the incision is subsequently planned. All techniques currently used employ ionizing radiation, at potentially high doses. In the investigator's experience, they find that due to the various factors which include the type of operating table or frame, the body habitus of the patient (in particular, greater degrees of thoracic kyphosis, and obesity), the inadequacy of the xray images to cover the entire rib cage and the presence of arms tucked to the side often make the localization process tedious and often leaves us with a certain degree of uncertainty.

Ultrasound has been used by various specialties, most notably by anaesthetists and pain specialties to perform point of care interventions to thoracic vertebrae. Ultrasound has also been used in the thoracic region to diagnose rib fractures. Counting the rib levels to localize the appropriate thoracic vertebral level was devised as a progression on these methods.

By showing that the use of ultrasound to count the ribs is a quick and accurate way to localize the appropriate spinal level, the need to expose patients to repeated doses of radiation can be eliminated.

The investigators hypothesize that the use of ultrasound will allow us to accurately determine the appropriate spinal level prior to the start of surgery by counting the ribs. This method will not only be precise, but it will also be quick, non-invasive, cheaper and will limit the amount of radiation that the patient is exposed to.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing thoracic spine surgery

Exclusion Criteria:

Paediatric patients or patients who are unable to give consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | This binary data will be collected during surgery
  To correlate with standard of care (fluoroscopy) - to ensure correct spinal levels marked on the skin

IPD SHARING:
Plan to Share IPD: No
No intention to share individual data